CLINICAL TRIAL: NCT03085862
Title: Lung Ultrasonography for Detecting Extravascular Lung Water Overload in Intensive Care Patients Early After Surgery: a Preliminary Study
Brief Title: Lung Ultrasonography and Extravascular Lung Water
Status: Completed | Type: Observational
Sponsor: General Hospital Sveti Duh (Other)
Responsible Party: Principal Investigator, Maja Karaman Ilic, Principal Investigator, General Hospital Sveti Duh
Other Study IDs: GHSvetiDuh
Record Dates: First submitted 2017-02-23; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Extravascular Lung Water
Keywords: Ultrasonography; Extravascular lung water; PaO2/FiO2 ratio

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung ultrasound and EVLW: This prospective study involved 60 patients without known cardiac or pulmonary diseases admitted to the intensive care unit at our hospital after elective abdominal or vascular surgery. The inferior vena cava collapsibility index (IVCcl), PaO2/FiO2 ratio, and appearance of B-lines ≤7 mm were determined upon admission to the intensive care unit and at 6, 12, and 24 h later. Fluid overload was defined as IVCcl ≤ 40% and the presence of B-lines ≤7 mm. Tissue oxygenation impairment was defined as a PaO2/FiO2 ratio < 200.

SUMMARY:
Aim. To investigate whether lung ultrasound can be used to detect extravascular lung water (EVLW) overload in the intensive care unit early after surgery.

Methods. This prospective study involved 60 patients without known cardiac or pulmonary diseases admitted to the intensive care unit at our hospital after elective abdominal or vascular surgery. The inferior vena cava collapsibility index (IVCcl), oxygen partial pressure (PaO2) and inspired oxygen pressure (FiO2) ratio (PaO2/FiO2), and appearance of B-lines ≤7 mm were determined upon admission to the intensive care unit and at 6, 12, and 24 h later. Fluid overload was defined as IVCcl ≤ 40% and the presence of B-lines ≤7 mm. Tissue oxygenation impairment was defined as a PaO2/FiO2 ratio < 200.

DETAILED DESCRIPTION:
After receiving general anesthesia, all patients received an endotracheal tube. After Co induction, anesthesia was maintained using a combination of inhalation anesthetic and intravenous drugs. Protective ventilation was combined with low flow. During surgery, all patients received Plasma Lyte 148 (pH 7.4; Viaflo, Baxter, Deerfield, IL, USA) at 6-8 ml/kg/h. Norepinephrine was administered at doses of 0.05-0.1 mcg/kg/min when needed to maintain mean arterial pressure over 60 mmHg. Packed red blood cells were used when hemoglobin concentration was ≤8.0 g/dl. At the end of anesthesia, participants were subjected to the recruitment maneuver. Patients older than 18 years admitted to intensive care unit after abdominal and vascular surgery with no cardiac or pulmonary diseases were included in the study.

.

After surgery, patients were admitted to the intensive care unit and given crystalloid Plasma Lyte at 1.5 ml/kg/h. At 24 h after surgery, all patients received the diuretic furosemide (20 mg).

Data on oxygen partial pressure and inspired oxygen pressure ratio (PaO2/FiO2), inferior vena cava collapsibility index (IVCcl) and occurrence of dense B-lines were monitored upon admission to the intensive care unit (baseline), as well as at 6, 12 and 24 h after admission. All measurements were done with the patients in supine position.

A decrease in PaO2/FiO2 ratio below 200 was taken to indicate a rise of extravascular lung water (EVLW) above 10 ml/kg (1-4); this cut-off indicates >20% shunting (5). IVCcl was measured based on changes in the diameter of the inferior vena cava during spontaneous breathing. IVCcl ≤40% was taken to indicate a rise in EVLW, since this cut-off reflects right arterial pressure of 10-15 mmHg (6). The appearance of "dense B-lines" on lung ultrasonography, defined as lines ≤7 mm apart, was also considered a sign of incipient increase in EVLW volume (7). Taking PaO2/FiO2 ratio as the reference method, we assessed the ability of dense B-lines, alone or in conjunction with IVCcl, to diagnose EVLW.

Statistical analysis was performed using SPSS 13 (Armonk, NY,USA). Independent-sample t tests were used to assess the significance of differences within groups for each set of measurements separately. The threshold of significance was p < 0.05. Possible correlation of PaO2/FiO2 ratio with occurrence of dense B-lines or with IVCcl ≤40% was assessed using the chi-squared test.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years admitted to the intensive care unit following elective abdominal or vascular surgery

Exclusion Criteria:

* known cardiac or pulmonary diseases
* lung ultrasonography showed unilateral distribution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years admitted to the intensive care unit at Clinical Hospital Sveti Duh (Zagreb, Croatia) following elective abdominal or vascular surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2015-11-20 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Inferior vena cava collapsibility index (IVCcl) | Baseline- upon admission to the ICU, 6, 12 and 24 hours after admission.
  The maximum and minimum IVC diameters (cm) were calculated using ultrasound. IVCcl was measured using formula [(maximum IVC diameter - minimum IVC diameter)/maximum IVC diameter] based on changes in the diameter of the inferior vena cava during spontaneous breathing. IVCcl ≤40% was taken to indicate a rise in EVLW, since this cut-off reflects right arterial pressure of 10-15 mmHg.
oxygen partial pressure (PaO2) and inspired oxygen pressure (FiO2) ratio | Baseline- upon admission to the ICU, 6, 12 and 24 hours after admission.
  PaO2/FiO2 ratio will be measured from the arterial blood. A decrease in P/F ratio below 200 was taken to indicate a rise of EVLW above 10 ml/kg; this cut-off indicates >20% shunting.
Dense B-lines | Baseline- upon admission to the ICU , 6, 12 and 24 hours after admission.
  The appearance of "dense B-lines" on lung ultrasonography, defined as lines ≤7 mm apart, was also considered a sign of incipient increase in EVLW volume

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berkowitz DM, Danai PA, Eaton S, Moss M, Martin GS. Accurate characterization of extravascular lung water in acute respiratory distress syndrome. Crit Care Med. 2008 Jun;36(6):1803-9. doi: 10.1097/CCM.0b013e3181743eeb. PMID 18496374
- [Background] Phillips CR, Chesnutt MS, Smith SM. Extravascular lung water in sepsis-associated acute respiratory distress syndrome: indexing with predicted body weight improves correlation with severity of illness and survival. Crit Care Med. 2008 Jan;36(1):69-73. doi: 10.1097/01.CCM.0000295314.01232.BE. PMID 18090369
- [Background] Craig TR, Duffy MJ, Shyamsundar M, McDowell C, McLaughlin B, Elborn JS, McAuley DF. Extravascular lung water indexed to predicted body weight is a novel predictor of intensive care unit mortality in patients with acute lung injury. Crit Care Med. 2010 Jan;38(1):114-20. doi: 10.1097/CCM.0b013e3181b43050. PMID 19789451
- [Background] Tagami T, Sawabe M, Kushimoto S, Marik PE, Mieno MN, Kawaguchi T, Kusakabe T, Tosa R, Yokota H, Fukuda Y. Quantitative diagnosis of diffuse alveolar damage using extravascular lung water. Crit Care Med. 2013 Sep;41(9):2144-50. doi: 10.1097/CCM.0b013e31828a4643. PMID 23760152
- [Background] Covelli HD, Nessan VJ, Tuttle WK 3rd. Oxygen derived variables in acute respiratory failure. Crit Care Med. 1983 Aug;11(8):646-9. doi: 10.1097/00003246-198308000-00012. PMID 6409506
- [Background] Zhao Z, Jiang L, Xi X, Jiang Q, Zhu B, Wang M, Xing J, Zhang D. Prognostic value of extravascular lung water assessed with lung ultrasound score by chest sonography in patients with acute respiratory distress syndrome. BMC Pulm Med. 2015 Aug 23;15:98. doi: 10.1186/s12890-015-0091-2. PMID 26298866
- [Background] Itobi E, Stroud M, Elia M. Impact of oedema on recovery after major abdominal surgery and potential value of multifrequency bioimpedance measurements. Br J Surg. 2006 Mar;93(3):354-61. doi: 10.1002/bjs.5259. PMID 16463271